CLINICAL TRIAL: NCT01689272
Title: Improving of Morphological,Clinical Biochemical and Instrumental Functional Reserve Estimation of Donor Kidney
Brief Title: Functional Reserve Estimation of Donor Kidney
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nazarbayev University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0111RK00337
Record Dates: First submitted 2012-09-17; First posted 2012-09-21 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: End-stage Renal Disease
Keywords: Kidney transplantation,functional status,survival.
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Kidney transplantation (Experimental): Kidney transplantation from alive relative donor.
  Interventions: Procedure: Kidney Transplantation from alive relative donor

INTERVENTIONS:
Procedure: Kidney Transplantation from alive relative donor — Donor kidney sampling, preservation, transport and transplantation

SUMMARY:
The purpose of the study:

* To estimate the role of morphological, clinical, biochemical and imaging studies at stages of kidney transplantation (medical therapy, explantation, preservation, transplantation).
* To improve the ways of preserving optimal functional parameters of renal transplants.

DETAILED DESCRIPTION:
Terminal chronic renal failure (ESRD) as a result of almost any chronic kidney disease develops due to progressive loss of nephrons. This state is characterized by a gradual deterioration of the functional abilities of not only the kidneys, but also the whole body. Currently, ESRD is among the first ten causes of mortality .

Transplantation of donor organs is the only radical treatment for various diseases of the terminal, for patients with a fatal prognosis.

Kidney transplantation has allowed not only save lives, but also to return to normal life, tens of thousands of people. Survival of renal transplant recipients is growing.

Despite the progress made in many clinics worldwide in recent years in the field of transplantation, kidney transplantation, does not settle the problem of reperfusion injury and the associated post-transplant dysfunction with the absence of clear indicators of morphological, clinical, biochemical and instrumental methods to assess functional reserve of organs that remain relevant and meaningful.

ELIGIBILITY:
Inclusion Criteria:

* recipients-patients with end-stage renal disease;
* donor healthy people without absolute contraindications to the kidney transplantation;
* donor and recipients who are both in the genetic and non-genetic related to each other.
* obligatory immunological compatibility by HLA-phenotyping provided that the donor and recipient are not relatives with each other;
* negative result of cross-match between donors and recipients;
* presence of pre-existing lymphotoxic antibodies in a recipient less than 50%;
* absence of standard absolute contraindications in a donor and in a recipient for surgeric intervention.

Age is 18-60 years.

Exclusion Criteria:

* patients with absolute contraindications to surgery: diseases of organs and systems having a threating risk to the life of donor and recipient during and after surgery;
* immunological incompatibility between donor and recipient;
* high level of pre-existing lymphotoxic antibodies in a recipient more than 50%, uncorrected by Therapy;
* donor age is under 18 and over 60 years;
* incapable persons;
* absence of a notarized consent form to kidney transplantation;
* presence of the active phase of viral infection with hepatitis B and C;
* positive results of blood tests for HIV/AIDS, syphilis;
* patients with severe concomitant pathology of kidneys, (or) heart and (or)liver.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Functional Reserve Estimation of Donor Kidney | for 12 months
  Graft survival is assessed on the following criteria:
  * The duration of the functioning graft
  * Clinical, laboratory and device functioning graft.
  * Morphological and histological study of the stages of transplantation (for withdrawal, before implantation) and the post-transplant period (with the threat of rejection.) Study of the blood recipient: Laboratory tests of blood recipient: biochemical analysis, the composition of the electrolyte, acid-base status, the level of immunosuppressants. Immunological typing for HLA-system. Cross-typing of donor and recipient, the level of pre-existing limfotsitotoksicheskih antibodies in the recipient.Patients survival.

SECONDARY OUTCOMES:
Clinical and Laboratory,Imaging Parameters | From 2 hours to 7 days
  * Intraoperational Macroscopic Description of signs of kidney ischemia: turgor, colour, consistency of transplanted kidney, pulse characteristics of renal artery.
  * Signs of graft rejection: increasing of temperature, blood pressure, the levels of waste products (blood creatinine, blood urea).

OTHER OUTCOMES:
Pre-Operative Patients Health Status: Donor and Recipient | For 1 week
  * Patient-donor health status.
  * Concomitant somatic pathology of a patient-recipient.
  * Time for Kidney transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Gani M Kuttymuratov, Phd, Principal Investigator — Advisor to the Board Chairman
Locations (1):
- Republican Scientific Center for Emergency Medicine, Astana, Kazakhstan